CLINICAL TRIAL: NCT03717766
Title: Application of New Technologies in the Resection of Intracranial Tumors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-TIC-2018-53
Record Dates: First submitted 2018-09-25; First posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Intracranial Neoplasm
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Intraaxial brain tumors that are tributary to surgical treatment. Prospective observational study of the use and effectiveness of intraoperative neuronavigation ultrasound, intraoperative tractography, intraoperative fluorescence, advanced neuronavigation and intraoperative neurophysiology in the resection of intracranial supratentorial tumors.
  Interventions: Device: intraoperative neuronavigation ultrasound, intraoperative tractography, intraoperative fluorescence, advanced neuronavigation and intraoperative neurophysiology

INTERVENTIONS:
Device: intraoperative neuronavigation ultrasound, intraoperative tractography, intraoperative fluorescence, advanced neuronavigation and intraoperative neurophysiology — 5-aminolevulinic acid (5-ALA) is a pro-drug that causes fluorescent protoporphyrins that accumulate in malignant gliomas. Fluorescence can be visualized during surgery by the use of a modified microscope, which helps the surgeon define the margins of the tumor.
  Neuro-navigated intraoperative ultrasound is an imaging technique that allows us to visualize intracranial lesions during surgery and correlate them with the image provided by the neuronavigator, obtaining a real-time view of the lesion and possible tumor remains.
  To achieve greater tumor resections without increasing the incidence of neurological deficits, the use of intraoperative neuromonitoring has been progressively implemented. This technology and specifically the brain mapping allows us to locate the functional areas of the brain and perform more aggressive resections with lower morbidity

SUMMARY:
Main Outcome: To assess the effectiveness of new intraoperative technologies in the resection of intracranial tumors.

Design: Prospective observational study.

Method: Prospective observational study of the use and effectiveness of intraoperative neuronavigation ultrasound, intraoperative tractography, intraoperative fluorescence, advanced neuronavigation and intraoperative neurophysiology in the resection of intracranial supratentorial tumors.

Number of patients: 70 - 100.

Duration of the study: 3 years.

Ethical considerations: The study will be carried out following the international ethical recommendations for medical research in humans. Before beginning the study, the Ethical Committee of the Hospital of Santa Creu i Sant Pau approved the study protocol. It is about the study of surgical techniques that we use in our usual clinical practice.

Fundings: There are no funding sources.

ELIGIBILITY:
Inclusion Criteria:

* intraaxial brain tumors that are tributary to surgical treatment.

Exclusion Criteria:

* extra-axial brain tumors.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intraaxial brain tumors that are tributary to surgical treatment.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of intracranial tumor resection | 3 years
  Effectiveness of new intraoperative technologies in the resection of intracranial tumors in terms of percentage of intracranial tumor resection and neurological deficit

IPD SHARING:
Plan to Share IPD: No